CLINICAL TRIAL: NCT00005083
Title: Defining Functional Tissue in Brain Tumors With Integrated Neuroimaging (Pilot Study)
Brief Title: Functional Magnetic Resonance Imaging and 1H-Nuclear Magnetic Resonance Spectroscopic Imaging in Treating Patients With Newly Diagnosed Brain Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CDR0000067692; UCLA-9712069; NCI-G00-1726
Record Dates: First submitted 2000-04-06; First posted 2003-12-16 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult anaplastic astrocytoma; adult myxopapillary ependymoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult pilocytic astrocytoma; adult subependymoma; adult ependymoblastoma; adult oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Astrocytoma; Ependymoma; Oligodendroglioma; Glioma; Glioma, Subependymal; Neuroectodermal Tumors, Primitive; Gliosarcoma | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: conventional surgery
Procedure: magnetic resonance imaging
Procedure: magnetic resonance spectroscopic imaging

SUMMARY:
RATIONALE: New imaging procedures, such as functional magnetic resonance imaging and 1H-nuclear magnetic resonance spectroscopic imaging, may improve the ability to detect the extent of cancer in the brain.

PURPOSE: Phase II trial to study the effectiveness of functional magnetic resonance imaging and 1H-nuclear magnetic resonance spectroscopic imaging in treating patients who have newly diagnosed brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the definable topospecific relationship between functional neuroactivation measured by functional magnetic resonance imaging (fMRI) and chemostructural tissue measurements made with 1H-nuclear magnetic resonance spectroscopic imaging (1H-NMRSI) in patients with newly diagnosed brain tumors situated in the vicinity of the brain's language and motor regions. II. Determine if clinical improvement correlates with stronger imaging signatures of neuroactivation on fMRI in this patient population. III. Determine if functional loss during tumor recurrence or progression correlates with increases in choline and decreases in N-acetylaspartate on 1H-NMRSI in regions that previously displayed activation on fMRI or in associated underlying white matter regions in these patients.

OUTLINE: Patients undergo preoperative functional magnetic resonance imaging (fMRI), 1H-nuclear magnetic resonance spectroscopic imaging (1H-NMRSI), and conventional contrast MRI over 2 hours followed by neurofunctional motor and/or language neurofunctional testing. Intraoperatively, patients undergo corticography consisting of awake language mapping and motor cortex stimulation. Patients undergo repeat imaging and neurofunctional evaluation at 2 weeks following surgery and prior to any radiotherapy or chemotherapy. Patients also undergo neurological and neuropsychological testing consisting of basic gait, motor coordination, reflexes, hand motor, tongue motor, and language evaluation to measure baseline, preoperative, and postoperative clinical status and outcomes. Patients are followed every 4 months for 1 year.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study over 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed brain tumor Neuroradiological and clinical evidence of probable glioma Lesion in close proximity to language and motor areas No prior resection

PATIENT CHARACTERISTICS: Age: 18 to 55 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No other medical or psychiatric disorder No contraindications to MRI scanning (e.g., metal implants, dental prostheses other than fillings, contrast allergies)

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 1998-03

CONTACTS AND LOCATIONS:
Overall Officials: Jeffry Alger, PhD, Study Chair — Jonsson Comprehensive Cancer Center